CLINICAL TRIAL: NCT06871670
Title: Knee Extensors Force Control in People With Chronic Obstructive Pulmonary Disease
Brief Title: Force Control in Chronic Obstructive Pulmonary Disease
Acronym: NEUROTIGUE F
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Université de Toulon (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-005
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Muscle; Force control; Non-linear; Variability; Isometric contractions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COPD: Patients with chronic obstructive pulmonary disease
  Interventions: Other: Submaximal isometric contractions of knee extensors
- Control participants: Healthy individuals
  Interventions: Other: Submaximal isometric contractions of knee extensors

INTERVENTIONS:
Other: Submaximal isometric contractions of knee extensors — Brief isometric contractions performed at 10, 20, 30, 40, 50 and 60% of maximal voluntary force in a random order.

SUMMARY:
Maximal muscle strength is one of the most commonly assessed neuromuscular parameters in people with COPD due to its accessibility and relevance for prescribing an appropriate workload for resistance training. However, maximal force production is very rarely necessary during daily activities which requires production of submaximal and precisely controlled forces. Despite growing research on motor impairments in COPD, very little attention has been given to the effect of this disease on force control. Therefore, this research aims to better understand the potential deficits in force control caused by COPD, through the use of advanced signal processing methods (i.e., nonlinear approaches). We hypothesized that force control would be reduced in people with COPD compared to healthy individuals, particularly at low force levels.

DETAILED DESCRIPTION:
This observational study is based on the analyses of data (force signals) recorded during the first visit of NEUROTIGUE study (NCT04028973).

Force signals were recorded during brief submaximal isometric contractions of the knee extensors performed by both COPD patients and healthy individuals. Each participant performed contractions at different intensity of his/her maximal muscle strength : 10, 20, 30, 40, 50 and 60%. Two contractions of approximately 6s duration were performed at each intensity by all participants. For a given intensity (e.g., 10%), both contractions were performed in a row but different intensities were accomplished in a random order.

Force control will be assess using a conjunction of parameters to provide a comprehensive understanding of force variability (e.g., coefficient of variation, non-linear approaches).

ELIGIBILITY:
Inclusion Criteria:

COPD patients :

* GOLD II - III or IV
* FEV1 <80% of predicted values
* Men and women aged 40 years and over
* French-speaking participant
* BMI <30 kg / m²
* Stable condition (i.e. without exacerbation) for more than 15 days
* Able to express their consent in writing prior to any participation in the study
* Affiliates or beneficiaries of a social security
* Minimum score of 26 on the MMSE questionnaire of 3 months or less

Healthy volunteers :

* Men and women aged 40 years and over
* French-speaking participant
* BMI <30 kg / m²
* No known chronic respiratory, cardiovascular, metabolic, renal or neuromuscular pathologies
* Able to express their consent in writing prior to any participation in the study
* Affiliates or beneficiaries of a social security
* Minimum score of 26 on the MMSE questionnaire of 3 months or less

For all participants :

-Subject who has not objected to the reuse of data collected

Exclusion Criteria:

COPD patients :

* Alcoholism, i.e. > 21 glasses a week for men and >14 glasses a week for women
* Psychiatric pathologies or antecedent of behavioral disorders
* Patients treated with oral or systemic corticosteroids (> 0.5 mg / kg / day for > 7 days)
* Contraindication to the application of a magnetic field (i.e. right hip arthroplasty, pelvic / abdominal surgeries)
* Severe vision or hearing problems not corrected
* Patient oxygen dependent
* Patients in exclusion period from another research protocol
* Pregnant women (known pregnancy) or lactating women
* Patient deprived of liberty by a judicial or administrative decision
* Patient subject to a legal protection measure or unable to express their consent
* Patient who is not sufficiently fluent in reading and understanding the French language to be able to consent to participate in the study
* Patient unable to follow study procedures and to respect visits throughout the study period
* Person with a medical history that, in the opinion of the investigator, could interfere with the results of the study
* Any condition that, in the opinion of the investigator, could increase and compromise the safety of the person in the event that he / she participates in the study
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the aims of the study

Healthy volunteers:

* Alcoholism, i.e. > 21 glasses a week for men and >14 glasses a week for women
* Psychiatric pathologies or antecedent of behavioral disorders
* Patients treated with oral or systemic corticosteroids (> 0.5 mg / kg / day for > 7 days)
* Contraindication to the application of a magnetic field (i.e. right hip arthroplasty, pelvic / abdominal surgeries)
* Severe vision or hearing problems not corrected
* Subjects in exclusion period from another research protocol
* Pregnant women (known pregnancy) or lactating women
* Regular physical activity with a frequency greater than 3 sessions per week
* Participant deprived of liberty by a judicial or administrative decision
* Participant subject to a legal protection measure or unable to express their consent
* Participant who is not sufficiently fluent in reading and understanding the French language to be able to consent to participate in the study
* Participant unable to follow study procedures and to respect visits throughout the study period
* Person with a medical history that, in the opinion of the investigator, could interfere with the results of the study
* Any condition that, in the opinion of the investigator, could increase and compromise the safety of the person in the event that he / she participates in the study
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the aims of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in NEUROTIGUE study (NCT04028973)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Difference of the coefficient of variation (CV) of force signal between COPD patients and healthy participants for different contraction intensities. | 10-min
  CV (%) is calculated as the ratio between standard deviation (SD) of force signal during muscle contraction and the mean produced force during the contraction.

SECONDARY OUTCOMES:
Difference of the root mean square error (RMSE) of force signal between COPD patients and healthy participants for different contraction intensities. | 10-min
  RMSE (%) is calculated as the absolute difference between the average produced force and the target force expressed as a percentage of the target.
Difference of Sample Entropy (SampEn) of force signal between COPD patients and healthy participants for different contraction intensities. | 10-min
  SampEn is a non-linear approach allowing to quantify the regularity of force signal.
Difference of Determinism (DET) from Recurrence Quantification Analysis (RQA) of force signal between COPD patients and healthy participants for different contraction intensities | 10-min
  DET from RQA represent another non-linear approach allowing to assess the regularity of force signal.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Vallier, MD, PHD, Study Director — Université de Toulon
Locations (1):
- Université de Toulon, laboratoires Laboratoire J-AP2S, Toulon, VAR, France

IPD SHARING:
Plan to Share IPD: Undecided